CLINICAL TRIAL: NCT03096691
Title: Use of Pessary in Case of Cervical Insufficiency and Short Cervix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Dilsad Herkiloglu, Principal Investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 058
Record Dates: First submitted 2017-03-25; First posted 2017-03-30 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Preterm Labor
Keywords: cervical pessary; preterm labor; Cervical insufficiency
MeSH Terms: conditions — Obstetric Labor, Premature; Uterine Cervical Incompetence

STUDY DESIGN:
Intervention Model Description: 100 pregnant women with a preterm delivery history and / or a cervical length of less than 25 mm will be included among the pregnancies between 16 and 24 weeks of gestation referred to obstetric and perinatology clinics. Information about the use of disease pessaries and treatment success in preventing premature birth of the pessary will be provided. Urine culture and cervical culture samples will be taken from both groups of patients. In the presence of infection, the patient's treatment will be planned and out of work. If no infection is detected and the patient agrees to use the pessary, the pessary will be used to prevent premature birth.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- short cervix group (Active Comparator): cervical pessary in group with first pregnancy or no preterm labor
  Interventions: Device: cervical pessary
- group with cervical insufficiency (Active Comparator): cervical pessary in group with multiple preterm labor
  Interventions: Device: cervical pessary

INTERVENTIONS:
Device: cervical pessary — Silicone rings known as arabin pessary are used to support the cervix in women with a sonographic short cervix.
  Other Names: arabin pessary

SUMMARY:
Prematurity is the most important cause of obstetric morbidity and mortality. Health centers and obstetricians are trying to reduce the preterm birth rate by taking into account the permanent effects of premature birth on human life in the early and long term.

The most effective solution of preterm delivery is to determine the patients entering the risk group and to prevent preterm labor by putting the correct diagnosis at the right time. Recently, there have been studies on the efficacy of pessary practice in preventing preterm birth, but with the positive results of these studies, there has been hope for early birth prevention as well as other treatments.

The aim of this study is; To assess the effectiveness of pessary use in patients with high risk for preterm labor and prophylactic cervical length less than 25 mm below 25 weeks and with a history of cervical insufficiency.

DETAILED DESCRIPTION:
The aim of this study is; To assess the effectiveness of pessary use in patients with high risk for preterm labor and prophylactic cervical length less than 25 mm below 25 weeks and with a history of cervical insufficiency.

100 pregnant women with a preterm delivery history and / or a cervical length of less than 25 mm will be included among the pregnancies between 16 and 24 weeks of gestation referred to obstetric and perinatology clinics. Information will be given about the success of treatment in the prevention of early birth of the pessary and the use of the disease pessary. Urine culture and cervical culture samples will be taken from both groups of patients. In the presence of infection, the patient's treatment will be planned and out of work. If no infection is detected and the patient agrees to use the pessary, the pessary will be used to prevent premature birth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cervical length of 25 mm> and a preterm labor history in the previous pregnancy

Exclusion Criteria:

* Patients with vaginal bleeding, with congenital anomalies, chorioamnionitis

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-03-30 (Estimated); Study Completion 2017-03-30 (Estimated)

PRIMARY OUTCOMES:
Preterm delivery | Less than 34 weeks gestation
  Spontaneous delivery before 34 completed weeks

CONTACTS AND LOCATIONS:
Overall Officials: dilsad herkiloglu, MD, Principal Investigator — Zeynep Kamil Maternity and Children's Hospital
Locations (1):
- Zeynep Kamil Maternity and Children's Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicolaides KH, Syngelaki A, Poon LC, Picciarelli G, Tul N, Zamprakou A, Skyfta E, Parra-Cordero M, Palma-Dias R, Rodriguez Calvo J. A Randomized Trial of a Cervical Pessary to Prevent Preterm Singleton Birth. N Engl J Med. 2016 Mar 17;374(11):1044-52. doi: 10.1056/NEJMoa1511014. PMID 26981934
- [Background] Goya M, Pratcorona L, Merced C, Rodo C, Valle L, Romero A, Juan M, Rodriguez A, Munoz B, Santacruz B, Bello-Munoz JC, Llurba E, Higueras T, Cabero L, Carreras E; Pesario Cervical para Evitar Prematuridad (PECEP) Trial Group. Cervical pessary in pregnant women with a short cervix (PECEP): an open-label randomised controlled trial. Lancet. 2012 May 12;379(9828):1800-6. doi: 10.1016/S0140-6736(12)60030-0. Epub 2012 Apr 3. PMID 22475493
- [Background] Dharan VB, Ludmir J. Alternative treatment for a short cervix: the cervical pessary. Semin Perinatol. 2009 Oct;33(5):338-42. doi: 10.1053/j.semperi.2009.06.008. PMID 19796732